CLINICAL TRIAL: NCT01714791
Title: Effect of Osteopathy on Pulmonary Function in Patients After Coronary Artery Bypass Graft Surgery: a Randomized Controlled Trial
Brief Title: Effects of Osteopathic Treatment on Pulmonary Function After Coronary Artery Bypass Graft Surgery
Acronym: OSTinCARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of new inclusions due to a significant change in surgery technique. An endoscopic a-traumatic coronary artery bypass (endo-ACAB) approach is now used.
Sponsor: Hartcentrum Hasselt (Other)
Responsible Party: Principal Investigator, Roncada Gert, Principal Investigator, Hartcentrum Hasselt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.07/cardio09.01
Record Dates: First submitted 2012-10-18; First posted 2012-10-26 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Mechanical Complication of Coronary Artery Bypass Graft; Respiratory Depression; Pain; Quality of Life
Keywords: Coronary Artery Bypass Graft; Osteopathic Medicine; Vital Capacity; Quality of Life; Cardiac rehabilitation
MeSH Terms: conditions — Respiratory Insufficiency; Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Patients following the outpatient cardiac rehabilitation program.
  Interventions: Other: Usual care
- Usual care and Osteopathic treatment (Experimental): Patients following the outpatient cardiac rehabilitation program and receiving osteopathic treatment.
  Interventions: Other: Usual care; Other: Osteopathic treatment

INTERVENTIONS:
Other: Usual care — Patients exercise at a heart rate corresponding to 65% of baseline Vo2peak. Each exercise training session takes 40-60 minutes. Exercise time is apportioned as follows: 42% on the treadmill, 33% on the circle ergometer and 25% on the arm cranking device. All patients exercise under close supervision 3 days per week for a total duration of 12 weeks.
  Other Names: Outpatient cardiac rehabilitation
Other: Osteopathic treatment — Patients receive 4 osteopathic treatments (OT). OT is performed in week 4, 5, 8 and 12 postoperative. Depending on what is found in the patient, treatments consist mostly of one or more of the following approaches:
  * Structural High Velocity Low Amplitude-techniques.
  * Muscle Energy Techniques.
  * General osteopathic mobilisations.
  * Functional techniques (Sutherland-, Jones-techniques,…) including inhibition techniques.
  * Fascia techniques.
  * Soft tissue- and connective tissue techniques.
  * Neurovisceral and neurolymphatic reflex techniques.
  * Fluidal techniques (lymphatic manipulative techniques,...).
  * Visceral manipulations.
  * Neurocranial and viscerocranial techniques.
  Arms: Usual care and Osteopathic treatment

SUMMARY:
The purpose of this study is to determine the short and long term effects of osteopathic treatment on pulmonary function, pain and quality of life in patients after coronary artery bypass graft (CABG) surgery. The study is a randomized controlled trial.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is performed worldwide. Several studies have found that there is a decrease in pulmonary function, loss of thoracic mobility and a high prevalence of chronic poststernotomy pain (CPSP) after CABG. So far there is no effective treatment for these conditions. The OstinCare study aims to investigate whether osteopathic treatment has an added value in the treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Planned Coronary Artery Bypass Graft (CABG) surgery at the Jessa Hospital Hasselt
* Planned Endoscopic Atraumatic Coronary Artery Bypass (endo ACAB) surgery at the Jessa Hospital
* Planned Minimal Invasive Aortic Valve Replacement (mini AVR) surgery at the Jessa Hospital

Exclusion Criteria:

* Thoracic surgery in the past
* Redo CABG
* Complications after CABG, requiring long-term (more than 6 days) admission to intensive care
* Pathologies of the lungs
* Pathologies of the heart, other than the coronary artery disease
* Surgery in the sub diaphragmatic region: epigastric region, left and right hypochondriac region.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in slow vital capacity (SVC) at 12 weeks. | preoperative (baseline) and 12 weeks postoperative
  A Slow Vital Capacity (SVC) test will be performed at each time point.

SECONDARY OUTCOMES:
Change from baseline in slow vital capacity (SVC) at 52 weeks. | preoperative (baseline) and 52 weeks postoperative
  A SVC test will be performed at each time point.
Change from baseline in McNew quality of life questionnaire at 12 weeks. | 3 weeks postoperative (baseline) and 12 weeks postoperative
  McNew questionnaire will be done at 3 and 12 weeks after surgery.
Change from baseline in McNew quality of life questionnaire at 52 weeks. | 3 weeks postoperative (baseline) and 52 weeks postoperative
  McNew questionnaire will be done at 3, 12 and 52 weeks after surgery.
Change in pain from baseline on Visual Analogue Scale (VAS) at 12 weeks postoperative. | 3 weeks postoperative (baseline) and 12 weeks postoperative
  Pain will be evaluated at 3 and 12 weeks after surgery.
Change in pain from baseline on VAS at 52 weeks postoperative. | 3 weeks postoperative (baseline) and 52 weeks postoperative
  Pain will be evaluated at 3, 12 and 52 weeks after surgery.
Change in thoracic stiffness from baseline on VAS at 12 weeks postoperative. | 3 weeks postoperative (baseline) and 12 weeks postoperative
  Thoracic stiffness will be evaluated at 3, 12 weeks after surgery.
Change in thoracic stiffness from baseline on VAS at 52 weeks postoperative. | 3 weeks postoperative (baseline) and 52 weeks postoperative
  Thoracic stiffness will be evaluated at 3, 12 and 52 weeks after surgery.

OTHER OUTCOMES:
Change from baseline in maximal aerobic capacity (VO2max) at 12 weeks postoperative | 3 weeks postoperative (baseline) and 12 weeks postoperative
  All patients will perform a maximal cardiopulmonary exercise test on a cycle ergometer. The test will be performed at the cardiac rehabilitation centre by a trained operator and under supervision of a cardiologist.
Changes in thoracic mobility at 4, 12 and 52 weeks postoperative. | 4, 12 and 52 weeks postoperative
  Osteopathic clinical examination of the thorax.

CONTACTS AND LOCATIONS:
Overall Officials: Gert Roncada, DO, MSc, Principal Investigator — Heart Centre Hasselt
Locations (1):
- Cardiac rehabilitation centre at the Jessa Hospital Hasselt, Hasselt, Limburg, Belgium

REFERENCES:
- [Background] Kristjansdottir A, Ragnarsdottir M, Hannesson P, Beck HJ, Torfason B. Chest wall motion and pulmonary function are more diminished following cardiac surgery when the internal mammary artery retractor is used. Scand Cardiovasc J. 2004 Dec;38(6):369-74. doi: 10.1080/14017430410016396. PMID 15804805
- [Background] Kristjansdottir A, Ragnarsdottir M, Hannesson P, Beck HJ, Torfason B. Respiratory movements are altered three months and one year following cardiac surgery. Scand Cardiovasc J. 2004 May;38(2):98-103. doi: 10.1080/14017430410028492. PMID 15204235
- [Background] Ragnarsdottir M, Kristinsdottir EK. Breathing movements and breathing patterns among healthy men and women 20-69 years of age. Reference values. Respiration. 2006;73(1):48-54. doi: 10.1159/000087456. Epub 2005 Aug 11. PMID 16106113
- [Background] Ragnarsdottir M, KristjAnsdottir A, Ingvarsdottir I, Hannesson P, Torfason B, Cahalin L. Short-term changes in pulmonary function and respiratory movements after cardiac surgery via median sternotomy. Scand Cardiovasc J. 2004 Mar;38(1):46-52. doi: 10.1080/14017430310016658. PMID 15204247
- [Background] Bruce J, Drury N, Poobalan AS, Jeffrey RR, Smith WC, Chambers WA. The prevalence of chronic chest and leg pain following cardiac surgery: a historical cohort study. Pain. 2003 Jul;104(1-2):265-73. doi: 10.1016/s0304-3959(03)00017-4. PMID 12855337
- [Background] Kalso E, Mennander S, Tasmuth T, Nilsson E. Chronic post-sternotomy pain. Acta Anaesthesiol Scand. 2001 Sep;45(8):935-9. doi: 10.1034/j.1399-6576.2001.450803.x. PMID 11576042
- [Background] Locke TJ, Griffiths TL, Mould H, Gibson GJ. Rib cage mechanics after median sternotomy. Thorax. 1990 Jun;45(6):465-8. doi: 10.1136/thx.45.6.465. PMID 2392792
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] Meyerson J, Thelin S, Gordh T, Karlsten R. The incidence of chronic post-sternotomy pain after cardiac surgery--a prospective study. Acta Anaesthesiol Scand. 2001 Sep;45(8):940-4. doi: 10.1034/j.1399-6576.2001.450804.x. PMID 11576043
- [Background] van Gulik L, Janssen LI, Ahlers SJ, Bruins P, Driessen AH, van Boven WJ, van Dongen EP, Knibbe CA. Risk factors for chronic thoracic pain after cardiac surgery via sternotomy. Eur J Cardiothorac Surg. 2011 Dec;40(6):1309-13. doi: 10.1016/j.ejcts.2011.03.039. Epub 2011 May 10. PMID 21561786
- [Background] van Leersum NJ, van Leersum RL, Verwey HF, Klautz RJ. Pain symptoms accompanying chronic poststernotomy pain: a pilot study. Pain Med. 2010 Nov;11(11):1628-34. doi: 10.1111/j.1526-4637.2010.00975.x. PMID 21044253
- [Background] Westerdahl E, Lindmark B, Bryngelsson I, Tenling A. Pulmonary function 4 months after coronary artery bypass graft surgery. Respir Med. 2003 Apr;97(4):317-22. doi: 10.1053/rmed.2002.1424. PMID 12693792
- [Background] Hansen D, Dendale P, Berger J, Meeusen R. Rehabilitation in cardiac patients:what do we know about training modalities? Sports Med. 2005;35(12):1063-84. doi: 10.2165/00007256-200535120-00005. PMID 16336009
- [Background] Alston RP, Pechon P. Dysaesthesia associated with sternotomy for heart surgery. Br J Anaesth. 2005 Aug;95(2):153-8. doi: 10.1093/bja/aei152. Epub 2005 May 13. PMID 15894562
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Derived] Roncada G. Osteopathic treatment leads to significantly greater reductions in chronic thoracic pain after CABG surgery: A randomised controlled trial. J Bodyw Mov Ther. 2020 Jul;24(3):202-211. doi: 10.1016/j.jbmt.2020.03.004. Epub 2020 Mar 17. PMID 32825989
- [Derived] Roncada G. Effects of osteopathic treatment on pulmonary function and chronic thoracic pain after coronary artery bypass graft surgery (OstinCaRe): study protocol for a randomised controlled trial. BMC Complement Altern Med. 2016 Nov 25;16(1):482. doi: 10.1186/s12906-016-1468-3. PMID 27884147